CLINICAL TRIAL: NCT02012972
Title: Non-Communicable Diseases and Antiretroviral Therapy Outcomes in the RapIT Study Population
Acronym: RapIT-NCD
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Collaborators: University of Witwatersrand, South Africa (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); City of Johannesburg (Unknown)
Responsible Party: Sponsor
Other Study IDs: H-32549; U01AI100015 (NIH); M130958 (Other: Wits University HREC (Medical))
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Antiretroviral Therapy, Highly Active; Diabetes Mellitus, Type 2; Cardiovascular Diseases
Keywords: Antiretroviral therapy; HIV/AIDS; Non-communicable diseases; South Africa
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Acquired Immunodeficiency Syndrome; Noncommunicable Diseases | interventions — Referral and Consultation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NCD Risks: Study subjects with NCD risks or disease at enrollment. Each of these subjects will have a Referral for NCD care
  Interventions: Behavioral: Referral for NCD care
- No NCD Risks: Study subjects without NCD risks or disease at enrollment.

INTERVENTIONS:
Behavioral: Referral for NCD care — Subjects in the NCD Risks group not already receiving care for the condition will be referred to a primary health clinic for care.
  Groups: NCD Risks

SUMMARY:
For national antiretroviral therapy (ART) programs, the most important health system goals in reducing morbidity and mortality among HIV-infection patients are to initiate treatment as early as eligibility criteria allow and to achieve the highest possible long-term retention of patients on ART. In South Africa, cohort data have consistently found high attrition among ART patients, with the combined cumulative outcomes of death and loss to follow up averaging 25-40% over the first five years after ART initiation. Like many other middle income countries, South Africa also faces very high rates of non-communicable diseases (NCDs) and NCD risks. Despite this, there are virtually no studies looking at interactions between ART and NCDs, and none that have considered the effect of NCDs and NCD risk factors on achieving the second health system goal mentioned above: long term retention on ART.

DETAILED DESCRIPTION:
The main RapIT study focuses on rapid initiation of ART, with short-term (6-month) attrition from treatment and viral suppression as the primary outcomes. In this supplemental study, we will evaluate the role of NCDs and NCD risk factors on long-term retention on ART, with outcomes including mortality, loss to follow up, viral suppression and immunologic improvement, and physical functioning, ability to perform normal daily activities, and economic productivity among patients already on ART. The study will enroll up to 400 adult patients already on ART for ≥ 12 months at the RapIT study site. At enrollment, consented subjects will be screened for elevated levels of several NCD risk factors including body mass index; glucose using HbA1c levels; blood pressure and cholesterol; as well as signs of abnormalities in hepatic, renal, and lung function. A medical history will be taken, and a questionnaire will gather information about chronic pain, alcohol use, smoking, physical functioning, ability to perform normal daily activities, and economic productivity. Referral for further NCD diagnosis and care will be offered as needed. Existing electronic medical records will be accessed to obtain retrospective data since ART initiation and to follow subjects prospectively for up to 24 months after the enrollment screening is completed. Six months after enrollment, subjects with NCDs or at high risk of NCDs will be re-screened at a routine ART medication pickup visit to assess uptake of referral and whether risks, conditions, or outcomes have changed. The study will help identify reasons for poor outcomes on ART and point to interventions that will help achieve the overall goals of the national ART program.

ELIGIBILITY:
Inclusion Criteria:

* Adult ART patients >35 years old.
* Initiated ART at least 12 months prior to study enrollment.
* Presenting at study clinic for a routine ART monitoring visit.

Exclusion Criteria:

* Pregnant or within first six months post-partum.
* Already enrolled in the RapIT study or another research study.
* Stated intention to transfer care to another location during the next 12 months.
* Not physically or emotionally able to participate in the study, in the opinion of the investigators.
* Not willing or able to provide written informed consent to participate in the study.
* Previously enrolled in the same study.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be non-pregnant adults who initiated antiretroviral therapy (ART) for HIV at least 12 months prior to study enrollment and are at least 35 years old. The age restriction will allow the study to focus on older patients who are at greater risk of NCDs. Pregnant women will be excluded because they face a different set of NCD risks directly related to pregnancy; women less than 6 months post-partum are also excluded to allow for the remaining effects of pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
NCDs and NCD risk factors in the study population by time on ART | Baseline
  The outcomes for primary objective 1 will be NCDs and NCD risk factors in the study population by time on ART, including diabetes, cardiovascular disease, respiratory conditions, hypertension, obesity, and behavioral risks such as smoking and alcohol use.

SECONDARY OUTCOMES:
HIV treatment outcomes | Baseline
  The outcomes for primary objective 2 will be HIV treatment outcomes, including all-cause mortality, loss to follow up (defined as having missed a scheduled medical or ART pick up visit by >90 days), attrition from ART care (defined as mortality or loss to follow up), viral suppression (defined as <400 copies/ml), physical functioning (as assessed by questionnaire) and economic productivity (also as assessed by questionnaire).
Uptake of NCD care | 6 months
  Uptake of non-communicable disease (NCD) care, defined as a patient newly diagnosed with an NCD or serious risk factor and referred for care who enroll for care at the study site or another clinic
Changes in NCD risks or prevalence | 6 months
  Changes in tests results or self-reported risks post-referral for those obtaining NCD care, defined by screening test results or questionnaire responses six months after referral to care

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Rosen, MPA, Principal Investigator — Boston University
Locations (1):
- Thuthukani Health Centre, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No